CLINICAL TRIAL: NCT06013189
Title: Re-Adjustment of Sweep Gas Flow to the During the Rewarming Period of the Cardiopulmonary Bypass to Prevent Alkalosis
Brief Title: Re-Adjustment of Sweep Gas Flow to the During the Rewarming Period of the Cardiopulmonary Bypass
Status: Recruiting | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Melis Tosun, Principal Investigator, Acıbadem Atunizade Hospital
Other Study IDs: ATADEK 2019-19/21
Record Dates: First submitted 2023-08-16; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Optimal Sweep Gas Flow; Determination of Optimal Sweep Gas Flow for Different Phases of Cardiopulmonary Bypass
Keywords: sweep gas flow; rewarming; cardiopulmonary bypass; alkalosis
MeSH Terms: conditions — Alkalosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Sweep Gas Flow did not changed (1.35 L/m2/min)
- Group 2: Sweep Gas Flow decreased during rewarming (1.2 L/m2/min)
  Interventions: Other: Gas Flow Adjustment
- Group 3: Sweep Gas Flow decreased during rewarming (1 L/m2/min)
  Interventions: Other: Gas Flow Adjustment

INTERVENTIONS:
Other: Gas Flow Adjustment — Decreased gas flow causes PaCO2 to elevate and prevents alkalosis
  Groups: Group 2; Group 3

SUMMARY:
The investigators designed this prospective observational study with the theory that alkalosis caused by decreased CO2 solubility due to temperature increase during the rewarming period of the Cardiopulmonary Bypass could be prevented by reducing the sweep gas flow during the rewarming period.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Elective CPB surgery

Exclusion Criteria:

* Patients undergoing minimally invasive surgery
* Patients undergoing robotic cardiac surgery,
* Patients undergoing deep hypothermia,
* Patients undergoing total circulatory arrest,
* Patients whose FiO2 requirement is high that cannot be applied to target gas flow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age scheduled for elective CPB surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
Arterial pH lever lower than 7.30 | during the cardiopulmonary bypass and postoperative 24th hour
  maintaining physiological pH

SECONDARY OUTCOMES:
rSO2 20% below initial value | during the cardiopulmonary bypass
  observing the rSO2 of brain during rewarming period

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Altunizade Hastanesi İstanbul, Istanbul, Altunizade, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No